CLINICAL TRIAL: NCT03322527
Title: Evaluation of the Technique LHP (Laser HemorrhoidoPlasty) in Haemorrhoidal Prolapse Mini Invasive Surgery Grade II or III of Goligher
Brief Title: Evaluation of the Technique LHP (Laser HemorrhoidoPlasty) in Haemorrhoidal Prolapse Mini Invasive Surgery
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: HLASER
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Hemorrhoids
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Hemorrhoids surgery technics evolved during the past 20 years. Recently a new one using laser have been developped. It aims at reducing the blood flow towards hemorroïdal plexuses by photocoagulating with a fiber laser the terminal branches of the superior rectal artery.

The aim is to evaluate the efficacy of this technic and note the post surgery pain and events

ELIGIBILITY:
Inclusion Criteria:

* age > 18
* hemorrhoid prolapse grade 2 and 3
* accepting participation

Exclusion Criteria:

* hemorrhoid prolapse grade 1 and 4
* other proctological pathology
* previous surgery of prolapsus
* with anti coagulant treatment
* Intestinal chronic inflammatory disease
* age < 18
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patient with a haemorroid proloapse surgery programmed in GHPSJ
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2016-12-19 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Goligher score | 1 year
  score evaluating symptoms of haemorroidal pathology

CONTACTS AND LOCATIONS:
Overall Officials: DE PARADES Vincent, MD, Principal Investigator — GHPSJ
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France